CLINICAL TRIAL: NCT01491750
Title: Factors Affecting Guided Imagery Response in Total Knee Replacement
Brief Title: Guided Imagery Response in Total Knee Replacement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kent State University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, ANN F JACOBSON, Professor, College of Nursing, Kent State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21AT003913-01A2 (NIH); R21AT003913-01A2 (NIH)
Record Dates: First submitted 2011-10-04; First posted 2011-12-14 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Osteoarthritis
Keywords: SURGERY; TOTAL JOINT REPLACEMENT; TOTAL KNEE REPLACEMENT; GUIDED IMAGERY; COMPLEMENTARY AND ALTERNATIVE THERAPY
MeSH Terms: conditions — Osteoarthritis | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GUIDED IMAGERY (Experimental)
  Interventions: Behavioral: GUIDED IMAGERY
- AUDIO BOOK (Placebo Comparator)
  Interventions: Behavioral: PLACEBO

INTERVENTIONS:
Behavioral: GUIDED IMAGERY — DAILY LISTENING TO A GUIDED IMAGERY CD FOR 2 WEEKS BEFORE AND 3 WEEKS AFTER SURGERY
  Arms: GUIDED IMAGERY
Behavioral: PLACEBO — DAILY LISTENING TO AN AUDIO BOOK SEGMENT FOR 2 WEEKS BEFORE AND 3 WEEKS AFTER SURGERY
  Arms: AUDIO BOOK

SUMMARY:
The purpose of this mixed methods pilot study is to produce preliminary data for a randomized, placebo-controlled trial testing a biobehavioral model of the effects of guided imagery on outcomes of total knee replacement surgery.

DETAILED DESCRIPTION:
The study uses a mixed-method design (quantitative experimental pilot study with qualitative descriptive and multiple case study methods) to address the study aims:

AIM 1: Generate estimates of effect sizes and assess feasibility of procedures for a future RCT testing a model of a standardized, prerecorded guided imagery intervention on functional outcomes of TKR.

AIM 2: Elucidate the GI responder mechanism through analysis of the effect of imaging ability and other potential moderators on guided imagery's effects on TKR outcomes.

AIM 3: Analyze the effect of guided imagery on outcome expectancy, psychological distress, rehabilitation commitment and neuroimmune activation as mediators on TKR functional outcomes.

AIM 4: Identify patients' perspectives related to receiving, and participating in a study of, guided imagery intervention for total knee replacement surgery (TKR).

DESIGN The proposed study is a modified sequential explanatory mixed methods design consisting of a Phase I RCT combined with a Phase II qualitative descriptive and case study. Mixed-methods research is an ideal strategy for rigorous development of interventions such as GI for further clinical testing. By systematically combining quantitative and qualitative approaches, the method is uniquely able to produce information for evaluating an intervention's context, its interactions with participant characteristics, and the link between the intervention and the outcomes. A variety of mixed methods designs have been developed, each with a different emphasis on (denoted as UPPER CASE LETTERS), and sequence of (denoted as order of listing), qualitative (qual) and quantitative (quan) approaches. The sequential explanatory design (QUAN/qual), which is primarily quantitatively oriented, uses qualitative methods to further describe and explain within- and between-subject variation on quantitative outcomes in experimental studies.

After the initial quantitative (QUAN) data collection and analysis, criterion sampling will be used to identify average and extreme cases on values of the quantitative outcome variables in treatment groups. Qualitative (qual) data collection and analysis of these cases can provide additional information about the application, operation, and outcome of the intervention beyond statistical findings, and test the validity of conceptual links between the intervention and outcome. Qualitative methods permit fuller exploration of subjective processes as they evolve during a major health care experience and uncover the complex and dynamic nature of these processes, and are particularly suited for gaining description and insight regarding responses to alternative therapies. The sequential explanatory method is thus well-suited for a study of the effects of a CAM intervention. The mixed method design also helps to clarify participants' views of the actual nature of an intervention, including the burden of treatment, and to reveal unanticipated situational constraints and enhancements to its execution.

METHODS In accord with the sequential explanatory design, the project will involve three phases: Phase I (QUAN): Quantitative data collection and analysis; Phase II (qual): Qualitative inquiry to amplify the quantitative findings; and Phase III: Final integration of findings to address the study aims and inform development of a subsequent RCT.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for a single TKR
* attendance at the hospital joint replacement class
* ability to speak, read, and write English -

Exclusion Criteria:

* current or planned use of guided imagery
* history of previous total joint replacement
* current enrollment in another clinical studY
* current treatment in a pain management program
* current diagnosis of immune disorders (e.g., rheumatoid arthritis, organ transplant, cancer, HIV, SLE)
* use of immune altering medications in past month
* comorbidities that would limit participation in study procedures or postoperative rehabilitation and/or impair recovery (e.g., psychosis; sensory, cognitive, neurologic or motor impairment
* vision or hearing deficits
* lymphedema
* morbid obesity [BMI > 40])
* reported diagnosis of anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
function | 6 months
  WOMAC AND SF-36

CONTACTS AND LOCATIONS:
Overall Officials: ANN F JACOBSON, PHD, Principal Investigator — Kent State University
Locations (1):
- Crystal Clinic Orthopaedic Center, Akron, Ohio, United States